CLINICAL TRIAL: NCT05931965
Title: Comparative Efficacy of Antidepressants With L-methylfolate, B12, and Magnesium in Depressive Disorders
Brief Title: Combination Therapy of Different Antidepressants With Dietary Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Riphah/IIMC/IRC/22/2069
Record Dates: First submitted 2023-06-14; First posted 2023-07-06 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Depression
Keywords: Depression; magnesium; Vit B12; L-methylfolate
MeSH Terms: conditions — Depression | interventions — 5-methyltetrahydrofolate; Vitamin B 12; mecobalamin; Magnesium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Antidepressant (No Intervention): Participants receive either escitalopram 10-20mg, sertraline 50-100mg, fluoxetine 20-40mg, duloxetine 30-60mg, mirtazapine 15-30mg, venlafaxine 75-150mg, trazodone 50-100mg, amitriptyline 25-75mg, or clomipramine 25-75mg orally daily for 4 weeks.
- Antidepressant and L-methylfolate (Experimental): Participants receive a combination of antidepressant and L-methylfolate 400µg twice daily orally for 4 weeks
  Interventions: Dietary Supplement: L-methylfolate
- Antidepressant and injectable mecobalamin (Experimental): Participants receive a combination of antidepressant and mecobalamin 500µg intramuscularly stat on alternate days (6 total injections)
  Interventions: Dietary Supplement: Vitamin B12
- Antidepressant and Magnesium (Experimental): Participants receive a combination of antidepressant and magnesium glycinate 400mg (Elemental: ≈120mg) twice daily orally for 4 weeks
  Interventions: Dietary Supplement: magnesium

INTERVENTIONS:
Dietary Supplement: L-methylfolate — Participants receive L-methylfolate 400µg orally twice daily for 4 weeks
  Other Names: 5-methyl-terahydrofolate
  Arms: Antidepressant and L-methylfolate
Dietary Supplement: Vitamin B12 — Participants receive mecobalamin 500µg intramuscularly stat on alternate days (6 total injections)
  Other Names: mecobalamin
  Arms: Antidepressant and injectable mecobalamin
Dietary Supplement: magnesium — Participants receive magnesium glycinate 400mg twice daily orally for 4 weeks (elemental 120mg approx.)
  Other Names: Mg
  Arms: Antidepressant and Magnesium

SUMMARY:
The aim of this clinical trial is to compare the effect of antidepressants in combination with different dietary supplements in patients with depression. Our main objective is to compare the efficacy of antidepressants in combination with either L-methyl folate, Vit B12, or magnesium) in patients with depressive disorders. The levels of depressive symptoms as measured by the Patient Health Questionnaire (PHQ-9) at base level and during follow-up.

DETAILED DESCRIPTION:
This is an open-label study assessing the comparative efficacy of antidepressants in combination therapy of either L-methylfolate, mecobalamin, or magnesium in patients with Depressive Disorder. The plan is to enroll 84 patients with depression based on Patient Health Questionnaire (PHQ-9) score of 9 and above, which is a valid and reliable Structured Clinical Interview. The investigators will collect data from the enrolled patient populations. The participants will be able to receive their results, on request, upon completion of the study. The investigators hypothesize that depressive symptoms can be improved by the addition of above mentioned nutritional supplementations with antidepressant medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Depressive Disorder having PHQ-9 Score 9 and above
* Age 12 and above
* Patients having low/marginal and low normal levels for arms 2 and 3 of respective supplements
* Patients having low/normal serum magnesium for arm 4

Exclusion Criteria:

* Patients having psychiatric diagnosis other than Depressive Disorder according to the International Classification of Diseases 11th Revision (ICD-11)
* History of kidney disease, myasthenia gravis
* Mentally handicapped or terminally ill patients
* Age less than 12 years
* Patients already taking multiple nutritional supplements
* Patients on polypharmacy with potential interactions with antidepressants and supplements in this study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Baseline and 4 weeks
  The change in the total PHQ-9 score between baseline and 4-weeks follow-up is the primary outcome measure. This measure is a patient-rated inventory of depressive symptoms. All items are scored on scales ranging from 0-3 and the sum of the scores provides the total score for the measure. On this scale, higher scores indicate poorer outcomes. Scores 9-19 and 20-27 are considered moderate and severe depression respectively.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Baseline, 2-weeks and 4-weeks
  The change in the total PHQ-9 score between baseline, and the intermediate 2-weeks, and 4-weeks follow-up is the secondary outcome measures. This measure is a patient-rated inventory of depressive symptoms. All items are scored on scales ranging from 0-3 and the sum of the scores provides the total score for the measure. On this scale, higher scores indicate poorer outcomes. Scores 9-19 and 20-27 are considered moderate and severe depression respectively.
Side-effects | Baseline, 2-weeks, and 4-weeks follow up
  A self-assessment questionnaire for undesirable effects in psychopharmacological treatment, developed by the Department of Psychiatry, Riphah International University, Pakistan. This is to investigate the presence or absence of 4 symptoms (diarrhea, drowsiness, insomnia, and rash), and their relationship with the treatment.
Depressive symptoms remission | Baseline, 2 weeks, 4 weeks
  Remission rate of Major Depression in the two groups over the course of treatment, defining remission as a score ≤ 4 on the PHQ-9 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Afifa Siddique, MBBS, Principal Investigator — IIMC-T, Riphah International University, Rawalpindi
Locations (1):
- Pakistan Railway Hospital, IIMC-T, Riphah International University, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serefko A, Szopa A, Poleszak E. Magnesium and depression. Magnes Res. 2016 Mar 1;29(3):112-119. doi: 10.1684/mrh.2016.0407. PMID 27910808
- [Background] Tarleton EK, Littenberg B, MacLean CD, Kennedy AG, Daley C. Role of magnesium supplementation in the treatment of depression: A randomized clinical trial. PLoS One. 2017 Jun 27;12(6):e0180067. doi: 10.1371/journal.pone.0180067. eCollection 2017. PMID 28654669
- [Background] Sun C, Wang R, Li Z, Zhang D. Dietary magnesium intake and risk of depression. J Affect Disord. 2019 Mar 1;246:627-632. doi: 10.1016/j.jad.2018.12.114. Epub 2018 Dec 27. PMID 30611059
- [Background] Noah L, Dye L, Bois De Fer B, Mazur A, Pickering G, Pouteau E. Effect of magnesium and vitamin B6 supplementation on mental health and quality of life in stressed healthy adults: Post-hoc analysis of a randomised controlled trial. Stress Health. 2021 Dec;37(5):1000-1009. doi: 10.1002/smi.3051. Epub 2021 May 6. PMID 33864354
- [Background] Chaban capital O, CyrillicS, Khaustova OO, Assonov DO, Sak LV. SAFETY AND EFFICACY OF THE COMPLEX DEPRILIUM(R) IN REDUCING SUBCLINICAL SYMPTOMS OF DEPRESSION IN PATIENTS WITH CHRONIC NON-COMMUNICABLE DISEASES: DOUBLE-BLIND RANDOMIZED CONTROLLED STUDY. Wiad Lek. 2023;76(1):136-144. doi: 10.36740/WLek202301119. PMID 36883502
- [Background] Maruf AA, Poweleit EA, Brown LC, Strawn JR, Bousman CA. Systematic Review and Meta-Analysis of L-Methylfolate Augmentation in Depressive Disorders. Pharmacopsychiatry. 2022 May;55(3):139-147. doi: 10.1055/a-1681-2047. Epub 2021 Nov 18. PMID 34794190
- [Background] Hardin A, Baldwin-Sayre C. L-Methylfolate as a Monotherapy for Treatment-Resistant Depression: A Case Study. Integr Med (Encinitas). 2020 Aug;19(4):14-18. PMID 33132780
- [Background] Dartois LL, Stutzman DL, Morrow M. L-methylfolate Augmentation to Antidepressants for Adolescents with Treatment-Resistant Depression: A Case Series. J Child Adolesc Psychopharmacol. 2019 Jun;29(5):386-391. doi: 10.1089/cap.2019.0006. Epub 2019 May 6. PMID 31058543
- [Background] Markun S, Gravestock I, Jager L, Rosemann T, Pichierri G, Burgstaller JM. Effects of Vitamin B12 Supplementation on Cognitive Function, Depressive Symptoms, and Fatigue: A Systematic Review, Meta-Analysis, and Meta-Regression. Nutrients. 2021 Mar 12;13(3):923. doi: 10.3390/nu13030923. PMID 33809274
- [Background] Carter B, Zenasni Z, Moat SJ, Hudson PR, Russell IT, McCaddon A; FolATED group consists of the following authors. Plasma Methylmalonic Acid Concentration in Folic Acid-Supplemented Depressed Patients with Low or Marginal Vitamin B-12: A Randomized Trial. J Nutr. 2021 Dec 3;151(12):3738-3745. doi: 10.1093/jn/nxab280. PMID 34510193
- [Derived] Siddique A, Khokhar MM, Waheed A, Naeem U, Aziz SA. Effect of combination therapy of methylfolate with antidepressants in patients with depressive disorder. BMC Pharmacol Toxicol. 2025 Jan 22;26(1):14. doi: 10.1186/s40360-025-00846-x. PMID 39844190